CLINICAL TRIAL: NCT05302882
Title: Evaluation of The Immediate Effect of Myofascial Release Application on Pain, Flexibility and Trunk Mobility in Patients With Chronic Low Back Pain
Brief Title: Evaluation of The Immediate Effect of Myofascial Release Application in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Ayşenur Çetinkaya, Lecturer, Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: acetinkaya
Record Dates: First submitted 2022-03-07; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Low-back Pain
Keywords: Myofascial release; Chronic low back pain; Flexibility
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Myofascial release was applied to the experimental group
  Interventions: Behavioral: Myofascial release
- Control Group (Active Comparator): Classical massage was applied to the control group
  Interventions: Behavioral: Classical massage

INTERVENTIONS:
Behavioral: Myofascial release — The physiotherapist placed both palms on the two right and left ribs at the T12 level and applied continuous stretching to the superior for 2 minutes. After this application, the physiotherapist placed one hand on the sacrum with the other hand on T12 with his hands crossed, and applied rhythmically 2 seconds of stretching and 2 seconds of relaxation for a total of 2 minutes. Then, myofascial release was terminated by applying deep compression to the paraspinal muscles with palms for 2 minutes on the right and 2 minutes on the left side, respectively.
  Arms: Experimental Group
Behavioral: Classical massage — Classical massage was applied to the lumbar region for 9 minutes. Classical massage was applied with the patient in the prone position. A small amount of solid vaseline was taken and a gentle stroke was applied for 1 minute to spread it sufficiently to the lumbar region. Then, superficial stroking was applied to the right paraspinal region for 1 minute from distal to proximal by the physiotherapist. After the same procedure was performed on the right paraspinal region for 1 minute. Then, both hands were placed on the right and left paraspinal region and friction was applied for 2 minutes. Afterwards, the patient's right paraspinal region was kneeding for 1 minute and then the same procedure was applied to the left paraspinal region for 1 minute. As the last procedure, the fingertips of both hands were placed on the right and left paraspinal region and the classical massage was completed by performing 2 minutes of deep euphlorage from the L5-S1 level to the T12 level.
  Arms: Control Group

SUMMARY:
Purpose: To determine the immediate effect of myofascial release application on pain, flexibility and trunk mobility in chronic low back pain (CLBP).

Materials and methods: Forty patients with CLBP participated in this experimental study. Participants were grouped in randomized control. Visual Analogue Scale (VAS) was used for pain assessment. Sit-Reach Test for flexibility evaluation and Straight Leg Raising Test with goniometric measurement for hamstring flexibility were used. Modified Schober Test was applied to evaluate trunk mobility. Comparison of the pre- and post-treatment evaluation data of the individuals in the same group was made using the "Wilcoxen Sum Rank Test", one of the non-parametric tests. Comparison of pre- and post-treatment evaluation data of both groups was performed using the non-parametric evaluation "Mann-Whitney U Test".

DETAILED DESCRIPTION:
It was aimed to determine the immediate effect of myofascial release application on pain, flexibility and trunk mobility in chronic low back pain (CLBP). Forty patients with CLBP participated in this experimental study. Participants were grouped in randomized control. Visual Analogue Scale (VAS) was used for pain assessment. Sit-Reach Test for flexibility evaluation and Straight Leg Raising Test with goniometric measurement for hamstring flexibility were used. Modified Schober Test was applied to evaluate trunk mobility. Comparison of the pre- and post-treatment evaluation data of the individuals in the same group was made using the "Wilcoxen Sum Rank Test", one of the non-parametric tests. Comparison of pre- and post-treatment evaluation data of both groups was performed using the non-parametric evaluation "Mann-Whitney U Test".

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 and 55 years;
2. low back pain lasting more than 3 months;
3. stable clinical status;
4. no cognitive and mental problems;
5. self-expression ability;
6. volunteering to participate in the study.

Exclusion Criteria:

1. problems of cooperation;
2. malignancy or infection;
3. acute fractures;
4. occlusive edema;
5. osteoporosis;
6. advanced degenerative joint problems;
7. acute rheumatologic conditions;
8. cortisone therapy;
9. use of blood thinners;
10. skin problems.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Pain Score | Baseline, immediately after the intervention
  The VAS is a widely used scale for pain assessment in daily practice. VAS, with 0-10 numbers on it and they are asked to give a value between these numbers. 0: I have no pain, 10: I have very severe pain
Change in The Straight Leg Raise Test Score | Baseline, immediately after the intervention
  test was used to assess hamstring flexibility. While the patient is in the supine position, the physiotherapist makes passive hip flexion with the knee straight and the measurement is made with a goniometer.
Change in The Modified Schober Test Score | Baseline, immediately after the intervention
  Test is an assessment method that measures lumbar flexion flexibility. The lumbosacral junction and 10 cm above were marked when the person was in an upright position. Then third mark was placed 5 cm below the lumbosacral junction. After anterior flexion as far forward as possible, the distance between the highest and lowest marks was measured.
Change in Sit and Reach Test Score | Baseline, immediately after the intervention
  test was used for flexibility evaluation. While the patient was performing maximum trunk flexion in the knee extension, the distance between the fingertip and the box aganist the sole of the foot was measured as +/- centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Halic University, Istanbul, Eyupsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boff TA, Pasinato F, Ben AJ, Bosmans JE, van Tulder M, Carregaro RL. Effectiveness of spinal manipulation and myofascial release compared with spinal manipulation alone on health-related outcomes in individuals with non-specific low back pain: randomized controlled trial. Physiotherapy. 2020 Jun;107:71-80. doi: 10.1016/j.physio.2019.11.002. Epub 2019 Nov 18. PMID 32026838
- [Result] Lohr C, Medina-Porqueres I. Immediate effects of myofascial release on neuromechanical characteristics in female and male patients with low back pain and healthy controls as assessed by tensiomyography. A controlled matched-pair study. Clin Biomech (Bristol). 2021 Apr;84:105351. doi: 10.1016/j.clinbiomech.2021.105351. Epub 2021 Apr 5. PMID 33848704
- [Result] Arguisuelas MD, Lison JF, Sanchez-Zuriaga D, Martinez-Hurtado I, Domenech-Fernandez J. Effects of Myofascial Release in Nonspecific Chronic Low Back Pain: A Randomized Clinical Trial. Spine (Phila Pa 1976). 2017 May 1;42(9):627-634. doi: 10.1097/BRS.0000000000001897. PMID 28441294